CLINICAL TRIAL: NCT05147519
Title: Multinational Observational Cohort of HIV and Other Infections (MOCHI)
Brief Title: Protocol RV 583 Multinational Observational Cohort of HIV and Other Infections
Acronym: MOCHI
Status: Recruiting | Type: Observational
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: RV 583; WRAIR # 2877 (Other: WRAIR)
Record Dates: First submitted 2021-11-02; First posted 2021-12-07 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
Keywords: STI; Observational
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Step 1: Step 1 will enroll participants aged 14-55 years who are vulnerable to contracting HIV. They will be evaluated every 12 weeks for HIV and other sexually transmitted infections (STIs).
  Interventions: Behavioral: Novel interventions to achieve HIV remission
- Step 2: Participants who are diagnosed with HIV will proceed to Step 2, with evaluation of viral load and other HIV-related tests every four weeks for 12 weeks and then every 12 weeks for a total of 48 weeks.
  Interventions: Behavioral: Novel interventions to achieve HIV remission
- Step 3: Participants who achieve and maintain viral suppression in Step 2 will proceed to Step 3 for continued HIV monitoring every 24 weeks to document maintenance of viral suppression and maintain engagement with the study site for potential future recruitment into interventional studies, including clinical trials of novel strategies to achieve HIV remission.
  Interventions: Behavioral: Novel interventions to achieve HIV remission

INTERVENTIONS:
Behavioral: Novel interventions to achieve HIV remission — To establish a group of well-characterized people living with HIV who initiated ART during acute or early HIV transmission that can serve as a source population for future studies, including those designed to test novel interventions to achieve HIV remission.

SUMMARY:
Multinational Observational Cohort of HIV and other Infections (MOCHI). This observational study is to gain information regarding the number of new HIV infections among people who engage in behaviors that make them vulnerable to acquiring HIV across multiple international sites.

DETAILED DESCRIPTION:
Prospective observational cohort study of participants vulnerable to HIV, conducted in three Steps. Step 1 will enroll participants aged 14-55 years who are vulnerable to contracting HIV. They will be evaluated every 12 weeks for HIV and other sexually transmitted infections (STIs). Participants who are diagnosed with HIV will proceed to Step 2, with evaluation of viral load and other HIV-related tests every four weeks for 12 weeks and then every 12 weeks for a total of 48 weeks. Participants who achieve and maintain viral suppression in Step 2 will proceed to Step 3 for continued HIV monitoring every 24 weeks to document maintenance of viral suppression and maintain engagement with the study site for potential future recruitment into interventional studies, including clinical trials of novel strategies to achieve HIV remission.

ELIGIBILITY:
Step 1 Inclusion Criteria Female or male aged 14-55 years Documented negative HIV test according to site-specific HIV testing procedures at entry/screening Able and willing to provide informed consent Willing to provide biometric identification Available for follow-up for the planned study duration Understands English or the local language as approved by the IRB, including people who are illiterate Willing to provide contact information for themselves and one personal contact who would know their whereabouts during the study period Willing to provide information regarding HIV risk behaviors and to undergo testing for HIV and other STIs

Considered to be vulnerable to HIV and other STIs based on any one or more of the following test results and/or self-reported behaviors:

1. Documented history of newly diagnosed syphilis, gonorrhea, chlamydia, Mycoplasma genitalium, herpes simplex virus, or acute hepatitis C virus infection in the 24 weeks prior to screening
2. Self-reported vaginal, oral, or anal intercourse in exchange for money as a regular source of income
3. Self-reported condomless vaginal or anal intercourse with at least three different partners living with HIV or of unknown status in the 24 weeks prior to screening
4. Self- reported injection drug use (IDU) in the 24 weeks prior to screening
5. Self-reported insertive or receptive anal or neovaginal intercourse with one or more different male or transgender partners in the 24 weeks prior to screening Step 1 Exclusion Criteria Any significant condition (medical, psychologic/psychiatric or social) that, in the judgment of the study investigator, might interfere with the conduct of the study Active drug or alcohol use or dependence that, in the judgement of the study investigator, would interfere with adherence to study requirements Current or past participation in a preventive or therapeutic HIV vaccine study, unless known placebo recipient Positive β-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) at screening for people of child-bearing potential and people who are amenorrheic for less than 12 consecutive months.

Step 2 Inclusion Criteria New diagnosis of HIV in the last 90 days during Step 1 as determined by site-specific HIV testing procedures Able and willing to continue follow-up for the planned study duration Step 2 Exclusion Criteria Any significant condition (medical, psychologic/psychiatric or social) that, in the judgment of the study investigator, might interfere with the conduct of the study Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements Step 3 Inclusion Criteria Virally-suppressed at the completion of Step 2 Adherent to ART Able and willing to continue follow-up for the planned study duration Step 3 Exclusion Criteria Any significant condition (medical, psychologic/psychiatric or social) that, in the judgment of the study investigator, might interfere with the conduct of the study Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The enrolled study population in step 1 will consist of up to 2500 men and women between 14 and 55 years of age who are vulnerable to HIV and other sexually transmitted infections. The incidence of HIV will be evaluated across all study sites as a primary objective; the incidence of STIs and retention in the cohort will be evaluated as key secondary objectives. During the accrual period, additional volunteers may be screened to replace participants lost to follow-up or withdrawn from the study, but no additional participants will be screened once the accrual period has expired.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Establish HIV Incidence at All Sites | 10 Years
  For the analysis of the incidence rate, only individuals who are not living with HIV at the baseline exam will be included in the incidence rate analysis.
  People without HIV will contribute person-time beginning with the time they enter the study until the study concludes or they are either censored or an HIV transmission event occurs. The event time for each subject is set to the minimum of the HIV transmission event time or the censoring time caused by one of the following: a drop-out event, a death event, or study end event. If one of these censoring events occurs, the censoring time is set to the last time there is recorded data for the subject. If an individual tests positive for HIV during the study, the HIV transmission event time is set to the visit during which the HIV transmission occurred. Those individuals who are lost to follow-up after enrollment will be censored at the last visit.

SECONDARY OUTCOMES:
Establish Incidence and Prevalence of STIs Including Chlamydia, Gonorrhea, Syphilis, and Mycoplasma genitalium | 10 Years
  For incident cases, the date of the positive test will be used as the date of infection. Specifically, for syphilis, a positive test can be determined by one of the following algorithms: 1. In the traditional algorithm, a non-treponemal test (e.g., rapid plasma reagin [RPR] or Venereal Disease Research Laboratory test [VDRL]) is used as the initial screen and reactive samples are confirmed with a treponemal test (e.g., fluorescent treponemal antibody absorption [FTA-ABS], T. pallidum particle agglutination [TPPA] test, Treponema pallidum particle agglutination assay [TPHA], or Syphilis IgG) or other tests that detect targets specific to T. pallidum. 2. The reverse algorithm uses a treponemal test for screening with reactive samples followed up with a non-treponemal test.
Willingness to Participate and Other Calculations | 10 Years
  Willingness to participate in an HIV vaccine trial and study retention rates and their respective 95% CIs will be estimated assuming a binomial distribution. Factors associated with willingness to participate in vaccine trial will be evaluated using logistic regression models. Self-reported risk behavior over time will be assessed by frequency tables and bar graphs. Changes in risk behavior over time will be evaluated using a Generalized Estimating Equation (GEE) model with clustering occurring within individuals (ex: multiple observations per person). Knowledge, attitudes, and practices regarding behaviors and preventive measures will be evaluated using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Trevor A. Crowell, MD, PhD, Principal Investigator — US Military HIV Research Program
Locations (3):
- Kenya Medical Research Institute/ USAMRD-A/Kenya (Kericho), Kericho, Kenya
- Institute of Clinical Epidemiology, National Institutes of Health, University of the Philippines Manila, Manila, Philippines
- Makerere University Walter Reed Program, Makerere, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No